CLINICAL TRIAL: NCT06945770
Title: Web-based Smoking Intervention as an add-on to Routine Smoking Cessation Clinical Treatment: a Randomized Controlled Trial
Brief Title: Web-based Smoking Intervention as an add-on to Routine Smoking Cessation Clinical Treatment
Acronym: POLSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, duygu altin, principal investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-4.1T/26; 29724 (Other Grant/Funding Number: EGE UNIVERSITY Office of Scientific Research Projects)
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
Keywords: tobacco use disorder; smoking cessation; web-based psycho-education
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — cytisine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POLSIS (Experimental): web based smoking cessation psycho-education
  Interventions: Behavioral: POLSIS; Drug: routine service delivery(Nicotine Replacement Theraphy, Cytisine)
- control (Active Comparator): routine service delivery
  Interventions: Drug: routine service delivery(Nicotine Replacement Theraphy, Cytisine)

INTERVENTIONS:
Behavioral: POLSIS — web based smoking cessation psycho-education
  Arms: POLSIS
Drug: routine service delivery(Nicotine Replacement Theraphy, Cytisine) — routine smoking cessation service delivery

SUMMARY:
This study evaluated the effectiveness of an online psycho-education program offered in addition to routine care for individuals attending a smoking cessation clinic. Conducted as a randomized controlled trial, the study assigned 103 participants to the intervention group and 105 to the control group. Based on follow-up data, analyses were carried out with 37 participants from the intervention group and 24 from the control group. Primary Hypotheses

Among individuals who applied to the Smoking Cessation Outpatient Clinic at the Institute on Drug Abuse, Toxicology, and Pharmaceutical Science, Ege University, those who receive additional online psychoeducational support integrated into the outpatient service are expected to:

H1: Be more successful in quitting smoking compared to those who do not receive this support.

H2: Be more successful in reducing the number of cigarettes smoked per day. H3: Show a significant change in their level of nicotine dependence.

Secondary Hypotheses H4: Show significant progress in the stages of change regarding smoking behavior.

H5: Show significant improvement in their mental well-being.

DETAILED DESCRIPTION:
Abstract Determination of Effectiveness of Online Psycho-education Embedded in Routine Service Delivery for Smoking Cessation: a Randomized Controlled Trial Objective: This study aims to evaluate the effectiveness of online psychoeducation provided in addition to routine treatment in a smoking cessation clinic compared to routine treatment alone.

Method: The study is a single-center, single-blind, randomized controlled experimental trial conducted between May 2024 and January 2025 at the Smoking Cessation Clinic of the Ege University Institute on Substance Abuse, Toxicology, and Pharmaceutical Sciences. Participants were randomly assigned to the intervention (n=103) and control (n=105) groups in a 1:1 ratio. During the study, the Warwick-Edinburgh Mental Well-being Scale Short Form (WEMWBS-SF), the Fagerström Nicotine Dependence Test (FNBT), and a case information form including HAPA stages of change were administered. The primary outcomes of this study are cigarette consumption, FNBT score, and smoking cessation success. The secondary outcomes include the HAPA stage of change and mental well-being score. Confounding variables considered in the study include education level, age, gender, employment status, mental health issues, marital status, and smoking cessation attempt. Based on follow-up data, analyses were conducted using data from 37 participants in the intervention group and 24 in the control group. Data analysis included paired and independent samples t-tests, chi-square analysis, one-way ANOVA, and linear and logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* using internet
* being a volunteer

Exclusion Criteria:

* not using internet
* not being a volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
the Fagerström Test for Nicotine Dependence (FTND) scores | from enrollment to the end of the treatment at 4 weeks
  Nicotine dependence was assessed using the Fagerström Test for Nicotine Dependence (FTND), a standardized scale ranging from 0 to 10, with higher scores indicating a greater level of nicotine dependence.
number of cigarettes smoked | from enrollment to the end of the treatment at 4 weeks
  number of cigarettes smoked on each day
smoking cessation | from enrollment to the end of the treatment at 4 weeks
  smoking less than 5 cigarettes

SECONDARY OUTCOMES:
mental well being score | from enrollment to the end of the treatment at 4 weeks
  The Short Form of the Warwick-Edinburgh Mental Well-Being Scale (SWEMWBS) consists of 7 items, each assessing positive feelings and thoughts experienced over the past two weeks. Participants rate how often they have experienced each statement during this period on a scale from 1 to 5 (1 = None of the time, 5 = All of the time). Higher scores indicate better mental well-being.
HAPA stage | from enrollment to the end of the treatment at 4 weeks
  HAPA stage of change (from 1 to 4)
  (1: I am not thinking about quitting smoking. 2:I am considering quitting smoking. 3:I am seriously thinking about quitting smoking. 4:I have already quit smoking.)

CONTACTS AND LOCATIONS:
Overall Officials: duygu altin, phd, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No